CLINICAL TRIAL: NCT00811161
Title: An Open Label Study to Evaluate the Efficacy of Airgent in Treating Damaged and Wrinkled Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PerfAction Ltd. (Industry)
Responsible Party: Dr. Dean D. AD-E/ Head, Department of Plastic Surgery & Burn Unit, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR12345
Record Dates: First submitted 2008-12-15; First posted 2008-12-18 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Wrinkles or Damaged Skin Condition
Keywords: Remodeling; Airgent; Hyaluronic acid; Collagen formation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- needle free injector of HA (Experimental)
  Interventions: Device: Airgent

INTERVENTIONS:
Device: Airgent — HA needle free injection, 3-4 treatments, 3-4 weeks apart

SUMMARY:
The primary objective of this study is to Evaluate the effectiveness of treatment of wrinkles or damaged skin with the Airgent device.

The secondary objective of this study are to:

* Evaluate subjects' satisfactory of the treatment.
* Demonstrate the safety of the Airgent treatment by evaluation of adverse events.

DETAILED DESCRIPTION:
Each subject will attend the clinic for the screening visit, 3 or 4 treatment visits 3-4 weeks apart, and number of follow-up visits (three at least). Evaluation of results of the performed treatments will be performed in course of the next treatment visit (prior to performance the next treatment) and at follow-up visits at 1, 3 and 6 months after the last treatment in session. Additional evaluation visits at 9 and 12 months after completion the treatment session can be performed upon decision of the investigator in case when considerable improvement is recorded during the 6-months evaluation visit.

Biopsies from up to five subjects treated for stretch marks will be collected at the time of 3-months evaluation visit, from treated and untreated zone (one of each).

Subjects will be requested to refrain from using any other method of skin rejuvenation for the entire duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Females and males in good general health 18-65 years old
* Subject that are capable of reading, following directions, and understanding the procedure to be applied and that are obligated to forgo any other method of skin rejuvenation treatment for the entire study period.

Exclusion Criteria:

* Medical or psychiatric conditions that can affect the subject's ability to give informed consent, or complete the study.
* Pregnant or lactating females.
* Other known diseases including diabetes, autoimmune disorders, epilepsy, severe migraines chronic liver or kidney
* Disease or contagious diseases, such as HIV or hepatitis
* Participation in a clinical trial within the last 30 days.
* Subjects on any medication (chronic use) that would affect the characteristic of the skin (medical or hormonal), such as NSAID, blood thinning medications, immunosuppressive drugs, steroids, vitamin E supplements and Isotretinoins within one month prior to enrollment.
* Subjects who have any form of suspicious lesion on the treatment area.
* Subjects with history of keloid formations or hypertrophic scarring.
* Subjects with permanent makeup/ tattoo (in the treated area).
* Subjects with any cutaneous inflammation on the treatment area such as herpes or acne.
* Subjects with known sensitivity to hyaluronic acid or to egg products.
* Subjects with clotting disorders.
* Subjects addicted to drug or alcohol.
* Subjects who underwent any aesthetic procedure in the treated area or adjacent to it.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Investigator/sub investigator assessment based on direct observation and photographs compared to baseline evaluation. | 3-12 months

SECONDARY OUTCOMES:
recording of adverse events. | 1-3 month
Evaluate subjects' satisfactory of the treatment | 1-12 month

CONTACTS AND LOCATIONS:
Overall Officials: Dean D. AD-EL D. AD-EL, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel